CLINICAL TRIAL: NCT03589872
Title: The Contribution of the Dual Task Interference on the Dexterity Related Activities of Daily Living in Parkinson's Disease
Brief Title: The Fine Motor Dexterity Under Dual Task in Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Sevim ACARÖZ CANDAN, Head of Department fo Physiotherapy and Rehabilitation, Ordu University
Other Study IDs: OrduU3
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Fine Motor Skill Dysfunction; Parkinson Disease
Keywords: hand function, dual task, Parkinson disease, activities of daily living
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: patients with parkinson disease
  Interventions: Diagnostic Test: Fine motor dexterity test, nine hole peg test

INTERVENTIONS:
Diagnostic Test: Fine motor dexterity test, nine hole peg test — The nine hole peg test will be performed under two different task (1)single task, (2)adding a cognitive task

SUMMARY:
This study was planned to investigate the contribution of dual task interference on dexterity related ADL disability in patients with Parkinson's disease. We hypothesised that the dual task interference is an indicator of dexterity related ADL difficulties.

DETAILED DESCRIPTION:
We planned this study as a cross sectional trial. 53 patients with Parkinson's disease will be evaluated under 2 different task by nine hole peg test. Besides this assessment the cardinal symptoms (bradykinesia, tremor, rigidity) will be evaluated to determine their contribution on the ADL performance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease according to the criteria of the United Kingdom brain Bank by neurologist
* Age 50-90 range
* having sufficient cognitive status according to the Mini Mental Status Evaluation (24 or above from the Mini Mental Test)

Exclusion Criteria:

* Having orthopedic and neurological disorders affecting hand function,
* Having sensory problems,
* Having Diabetus mellitus

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample:community-dwelling patients with Parkinson disease.
Sampling Method: Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
Nine hole peg test | 5 minutes
  The Nine-Hole Peg Test is used to measure finger dexterity in patients with various neurological diagnoses. The patient must pick up the pegs from the holes and replace them back as fast as possible. The Nine Hole Peg Test should be conducted with the dominant arm first, then nondominant hand. The time will be recorded in second to complete the test. The test will be performed under three task;
  1. single task: Only nine-hole peg test
  2. adding a cognitive task: Nine-hole peg test will be performed with a concurrent cognitive task. The cognitive task is a serial 7 subtraction from numbers changed between 290 and 310 during the performing nine-hole peg test. The time will be recorded.
ADL-related dexterity Questionnaire 24 (DextQ-24) | 10 minutes
  Dexterity-related ADL difficulties were measured by the ADL-related dexterity Questionnaire 24 (DextQ-24), including 24 question dealing with bimanual and unimanual activities, which is a reliable and valid disease specific questionnaire to evaluate dexterity in patients with PD. Each question is scored between 1 (no problems) and 4 (need aid to perform task) by the patient's experience. Total score ranged from 24 points to 96 points.

SECONDARY OUTCOMES:
Modified Hoehn and Yahr Scale | 2 minutes
  Disease progression will be assessed with modified Hoehn and Yahr Scale. The original scale included stages 1 through 5. Since then, stage 0 has been added, and stages 1.5 and 2.5 have been proposed. This modified scale allocates stages from 0 to 5 to indicate the relative level of disability.
  Stage 0: No signs of disease.
  Stage 1: Unilateral symptoms only.
  Stage 1.5: Unilateral and axial involvement.
  Stage 2: Bilateral symptoms. No impairment of balance.
  Stage 2.5: Mild bilateral disease with recovery on pull test.
  Stage 3: Balance impairment. Mild to moderate disease. Physically independent.
  Stage 4: Severe disability, but still able to walk or stand unassisted.
  Stage 5: Needing a wheelchair or bedridden unless assisted.
Unified Parkinson's Disease Rating Scale (UPDRS) - Section of Activities of Daily Living (ADL) | 10 minutes
  The UPDRS- ADL section evaluates the impact of Parkinson disease on ADL according to patient's perspective. The ADL section consists of 13 items for gathering information on the patient's own perception of functional impairment due to PD. Each item scores between 0-4. 0 means normal and 4 means severe impairment. The total score change between 0-52. High scores indicate severe impairment.
Unified Parkinson's Disease Rating Scale (UPDRS) - Motor Section | 10 minutes
  Motor section of UPDRS determines the impairment due to the Parkinson's disease. Rigidity, bradykinesia and tremor items which are relating with upper extremity function will be assessed. Each item scores between 0-4. 0 means normal and 4 means severe impairment. The total scores of rigidity, bradykinesia, and tremor, respectively range between 0-8, 0-24 and 0-16.

CONTACTS AND LOCATIONS:
Overall Officials: SEVİM ACARÖZ CANDAN, Principal Investigator — Ordu University, Department of Physiotherapy and Rehabilitation
Locations (1):
- Sevim ACARÖZ CANDAN, Ordu, Altinordu, Turkey (Türkiye)